CLINICAL TRIAL: NCT04870957
Title: University of Michigan Mechanistic Research Center -The Back Pain Consortium Research Program
Brief Title: The Back Pain Consortium Research Program Study
Acronym: BACPAC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Afton Hassett, Psy.D., Associate Professor of Anesthesiology, University of Michigan
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00180994; 1U19AR076734-01 (NIH)
Record Dates: First submitted 2021-04-28; First posted 2021-05-04 (Actual); Results first posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-10

CONDITIONS: Chronic Low-back Pain
Keywords: Pain; Back Pain
MeSH Terms: conditions — Pain; Back Pain | interventions — Exercise; Duloxetine Hydrochloride

STUDY DESIGN:
Intervention Model Description: Sequential, multiple assignment, randomized trial (SMART) design
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- MBSR (mindfulness-based stress reduction) (Experimental): Participants receiving MBSR during Treatment 1 or 2.
  Interventions: Behavioral: MBSR; Device: Pro-Diary monitor
- PT and exercise (Experimental): Participants receiving PT during Treatment 1 or 2.
  Interventions: Behavioral: PT and exercise; Device: Pro-Diary monitor
- Acupressure (Experimental): Participants receiving Acupresure during Treatment 1 or 2.
  Interventions: Device: Self -administered acupressure; Device: Pro-Diary monitor
- Duloxetine (Experimental): Participants receiving Duloxetine during Treatment 1 or 2.
  Interventions: Drug: Duloxetine; Device: Pro-Diary monitor
- Run-In (Experimental): Pre-treatment run-in period with access to the PainGuide self management platform.
  Interventions: Behavioral: PainGuide; Device: Pro-Diary monitor
- Follow-Up (No Intervention): Participants on Follow-Up at any timepoint throughout the study.

INTERVENTIONS:
Behavioral: PainGuide — A 4-week, online, self-management program for pain known as PainGuide (online or smart phone). Participants will use this during the run-in period as well as after the run-in period.
  Arms: Run-In
Behavioral: MBSR — In this group (mindfulness-based stress reduction) participants will take part in 9 group sessions.
  The groups sessions will be divided into 8 weekly 2-hour groups sessions and one 6-hour "retreat". During the sessions participants will practice mindfulness exercises directed by the a MBSR therapist. Additionally, participants will also be asked to practice daily formal mindfulness at home using audio recordings of 30-45 minute guided meditation exercises. These audio recordings can be accessed online. The sessions may take place in-person or virtually.
  Arms: MBSR (mindfulness-based stress reduction)
Behavioral: PT and exercise — Participants will take part in 10 physical therapy visits over the course of 8 weeks. Participants will meet with the physical therapist twice a week for a 1-hour session for weeks 1 and 2 and then weekly for the remaining 6 weeks. The physical therapist will tailor a program to the participant's needs according to recommended PT practice guidelines that will include in-person treatment, home exercise prescription, and encouragement of progressive, low-intensity, submaximal fitness and endurance activities, such as walking.
  Participants will be given a home program of exercises to be done daily and asked to engage in daily walking with a set goal based on the individual's capacity and current fitness level. Walking was selected as the aerobic exercise of focus for this treatment because it is recommended for patients with all levels of pain severity, is highly feasible to complete, and has shown effects on outcomes such as pain and disability.
  Arms: PT and exercise
Device: Self -administered acupressure — A device called the "AcuWand" will be used to administer the self-acupressure intervention for approximately 30 minutes daily for 8 weeks. Participants will use a mobile application (app) called "MeTime" that will have daily instructions on how to use the AcuWand. Research staff will show participants how to use the AcuWand and MeTime app. In addition, participants will keep a daily log to track at-home acupressure sessions.
  Arms: Acupressure
Drug: Duloxetine — For days 1-7, patients will take 30mg of duloxetine once a day, in the morning. Starting day 8, participants tolerating the medication will be escalated to 60mg once a day. They will also have the option of staying at 30mg, once a day or stopping the medication. At the end of the 8-week intervention period, participants will have the option to continue the medication commercially (non-study medication) under the care of their physician or taper off the medication. During the entire 8-week intervention, patients will be asked to keep a daily log of medication dosage, any missed doses, and any side-effects they may have experienced.
  Other Names: Cymbalta
  Arms: Duloxetine
Device: Pro-Diary monitor — Participants will wear during 5 separate 7-day "home monitoring" periods to assess physical activity (objectively measured via accelerometry), and ecological momentary assessment (EMA) of mental and physical symptoms. EMA will be collected during Weeks 1, 6, 15, 24 and 36.
  Other Names: Electronic wrist device that looks like a watch
  Arms: Acupressure; Duloxetine; MBSR (mindfulness-based stress reduction); PT and exercise; Run-In

SUMMARY:
This study is being completed to better understand who benefits from different chronic pain treatments and how these treatments work.

This study will include a four week run-in period for all cLBP participants. After completing the PainGuide (online or smart phone accessible website) run-in period, participants will be assessed using either the light or light plus deep phenotyping assessment battery and those who minimal or modest improvement in their pain (based on PGIC) will be randomized to one of four 8-week treatments (mindfulness-based stress reduction (MBSR), physical therapy (PT) and exercise, acupressure self-management, or duloxetine).

In addition, participants will complete study visits including physical exams, complete surveys, provide samples (blood,saliva, etc.), wear an electronic wrist device at certain times, and have Magnetic resonance imaging (MRIs) during the study.

Following one of the 4 treatments (8 weeks) if participants have a certain level of pain (that meets eligibility for more treatment) they will be then randomized to complete one of the 3 treatments that was not already assigned to them.

The study hypothesizes the following:

that this interventional response phenotyping can identify individuals with different underlying mechanisms for their pain who thus respond differentially to evidence-based interventions for chronic lower back pain (cLBP).

DETAILED DESCRIPTION:
In addition, the following mechanistic hypothesis and Aims are included:

Mindfulness-Based Stress Reduction:

Aim 2: the study predicts that patients with chronic low back pain (cLBP) will preferentially respond to this therapy if PROs indicate higher levels of pain catastrophizing, as measured by the Pain Catastrophizing Scale, or lower scores on the Experiences Questionnaire.

Aim 3: the study hypothesizes that cLBP patients with decreased activation in response to pain in the subgenual anterior cingulate cortex (sgACC) and Prefrontal Cortex and increased activation in somatosensory cortex (S1) and thalamus will respond preferentially to MBSR.

Physical Therapy (PT) and Exercise

Aim 2: The primary hypothesis for the light phenotyping protocol is those individuals with the highest scores on the Fear Avoidance Beliefs Questionnaire and lowest scores for PROMIS Self-Efficacy for Managing Symptoms will be most likely to improve from PT/Exercise program.

Aim 3: the study hypothesis that low vagal tone and high basal inflammation will predict responsiveness to the PT/Exercise program.

Acupressure:

Aim 2: The study hypothesizes that females with cLBP will respond better to acupressure than men, as will those with higher scores on the 2011 Fibromyalgia Survey Questionnaire.

Aim 3: The study predicts that cLBP patients with higher posterior insula glutamate and/or greater insula - Default Mode Network (DMN) connectivity (as well as increased DMN-S1 connectivity

Duloxetine:

Aim 2: the study hypothesizes that it will replicate previous studies suggesting that participants with cLBP will preferentially respond to this therapy if patient reported outcomes indicate stronger elements of either neuropathic pain (indicated by a high PainDETECT score) or centralized/nociplastic pain (indicated by more widespread pain on the 2011 Fibromyalgia Survey Questionnaire).

Aim 3: the study anticipates then that deficient pain inhibition on quantitative sensory testing, decreased periaqueductal gray (PAG)-insula connectivity, and elevated stimulated inflammatory responses will be associated with a positive response to centrally-acting duloxetine.

Additionally, a subset of individuals (n=160) from these groups will be asked to participate in an expanded phenotyping study that will include structural and functional brain neuroimaging, quantitative sensory testing (QST), plasma measures of inflammation, and digital measurement of autonomic tone.

ELIGIBILITY:
Inclusion Criteria for Light Phenotyping (all participants):

* Definition of cLBP described in the NIH Task Force Report on Research Standards for Chronic Low Back Pain (for example (i.e.), low back pain present at least six months, and present more than half of those days.
* Individuals must have the eligible protocol pain interference score on PROMIS Pain Interference.
* Individuals must be willing to be randomized to receive any of the four proposed treatments.

Exclusion Criteria for Light Phenotyping (all participants):

* History of discitis osteomyelitis (spine infection) or spine tumor
* History of ankylosing spondylitis, rheumatoid arthritis, polymyalgia rheumatica, or psoriatic arthritis, lupus
* History of cauda equina syndrome or spinal radiculopathy with functional motor deficit (strength <4/5 on manual motor testing)
* Diagnosis of any vertebral fracture in the last 6 months
* Osteoporosis requiring treatment other than vitamin D and calcium supplements
* Cancer (History of any bone-related cancer or cancer that metastasized to the bone, Currently in treatment for any cancer or plan to start cancer treatment in the next 12 months, History of any cancer treatment in the last 24 months)
* Life expectancy less than 2 years
* Unable to speak and write English
* Visual or hearing difficulties that would preclude participation
* Presence of any history that would preclude scanning in magnetic resonance imaging (MRI)
* Uncontrolled drug/alcohol addiction
* Individuals receiving disability or compensation within the past year, or involved in litigation
* Pregnancy or breastfeeding
* History of allergy to duloxetine
* Individuals on high doses of opioids (over 100 oral morphine equivalents (OME) per day)
* Scheduled back surgery, back surgery within the last year, or more than one back surgery in the past.
* Expecting to receive an injection of surgical procedure within the next year for their cLBP
* Current/planned (in the next 2 years) enrollment in another study of a device or investigational drug that would interfere with this study, this may include participation in a blinded trial.
* Any other diseases or conditions that would make a patient unsuitable for study participation as determined by the site principal investigators. This would include but not be limited to severe psychiatric disorders, active suicidal ideations or history of suicide attempts, and an uncontrolled drug and/or alcohol addiction

Contraindications to Study Intervention: duloxetine

* certain medications (per protocol)
* renal dysfunction (creatinine clearance <30 milliliters per minute (mL/min) or End- Stage Renal Failure)
* Hepatic dysfunction: Liver function tests (LFTs) elevated times 1.5

Contraindications to Study Intervention: Acupressure

* Currently receiving acupressure or acupuncture through formal therapy

Contraindications to Study Intervention: MBSR

* Current participation in a structured MBSR program

Contraindications to Study Intervention: PT & Exercise

* Currently receiving any type of structured manual therapy or exercise treatment for low-back pain.
* Contraindication for manual therapy and/or participation in an exercise program

Inclusion Criteria for Deep Phenotyping (subset 160 participants):

* Right hand dominant (such as the hand used when writing or throwing/catching a ball)
* Normal visual acuity or correctable (with corrective lenses- glasses or contacts) to at least 20/40 for reading instructions in the MRI and visual sensitivity testing
* No contraindications to MRI (i.e., metal implants)
* Willingness to refrain from taking any "as needed" medications, including pain medications such as Nonsteroidal anti-inflammatory drugs (i.e., Motrin, Advil, Aleve), acetaminophen, and opioids, for 8 hours before undergoing neuroimaging and 10.1 Quantitative Sensory Testing (QST)
* Willingness to refrain from alcohol and nicotine on the day of QST and neuroimaging (alcohol and nicotine consumption is allowed after testing is completed)
* Willingness to refrain from any unusual physical activity or exercise that would cause muscle and/or joint soreness for 48 hours prior to testing (routine exercise or activity that does not lead to soreness is acceptable)
* Able to lie still on back for 2 hours during MRI

Exclusion Criteria for Deep Phenotyping (subset 160 participants):

* Severe claustrophobia precluding MRI and evoked pain testing during scanning
* Diagnosed peripheral neuropathy
* Current, recent (within the last 6 months), or habitual use of artificial nails or nail enhancements. (Artificial nails can influence pressure pain sensitivity at the thumbnail)
* Body Mass Index greater than 45 or unable to comfortably fit in the bore of the MRI magnet

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2025-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Afton Hassett, PsyD, Principal Investigator — University of Michigan; Daniel Clauw, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Data (including bio-specimens, omic data, raw imaging data, and other study data) will be shared with consortial partners. Data will be held at a Data Acquisition Center (DAC) hosted at the University of North Carolina. Omics data will be shared through NIH portals as required. Data dictionaries are harmonized across study sites and shared with consortial partners.
Supporting Information: Study Protocol, ICF
Time Frame: Per the study data sharing plan, data will be shared to the consortial DAC at fixed intervals after 20% completion is attained (and then at each subsequent 20%). The consortium currently plans for perpetual access for consortial partners.
Access Criteria: The data will be available only to members of the consortium and is governed by a consortial data use agreement. Members must submit a request form for data access. The Data Access and Publications Committee will review requests and notify Data Access Team when access can be granted.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from June 1, 2021-June 27, 2024, through Michigan Medicine clinics (Back & Pain Center, Physical Medicine, Family Medicine, Neurosurgery) and community/online sources (UMHealthResearch.org, Facebook, MLive, flyers, radio). Of 6,965 screened, 494 eligible participants completed a baseline visit.
Pre-assignment Details: Participants completed a 4-week online PainGuide run-in before randomization. At T2, those with PGIC ≥ 2 were randomized to one of four 8-week treatments (MBSR, PT/exercise, acupressure, or duloxetine). Participants with PGIC < 2 entered follow-up only and were not randomized. Screen failures were those who did not meet eligibility criteria were withdrawn from the study.
Groups:
- MBSR (mindfulness-based stress reduction): MBSR: In this group (mindfulness-based stress reduction) participants will take part in 9 group sessions.
  The groups sessions will be divided into 8 weekly 2-hour groups sessions and one 6-hour "retreat". During the sessions participants will practice mindfulness exercises directed by the a MBSR therapist. Additionally, participants will also be asked to practice daily formal mindfulness at home using audio recordings of 30-45 minute guided meditation exercises. These audio recordings can be accessed online. The sessions may take place in-person or virtually.
  Pro-Diary monitor: Participants will wear during 5 separate 7-day "home monitoring" periods to assess physical activity (objectively measured via accelerometry), and ecological momentary assessment (EMA) of mental and physical symptoms. EMA will be collected during Weeks 1, 6, 15, 24 and 36.
- PT and exercise: PT and exercise: Participants will take part in 10 physical therapy visits over the course of 8 weeks. Participants will meet with the physical therapist twice a week for a 1-hour session for weeks 1 and 2 and then weekly for the remaining 6 weeks. The physical therapist will tailor a program to the participant's needs according to recommended PT practice guidelines that will include in-person treatment, home exercise prescription, and encouragement of progressive, low-intensity, submaximal fitness and endurance activities, such as walking.
  Participants will be given a home program of exercises to be done daily and asked to engage in daily walking with a set goal based on the individual's capacity and current fitness level. Walking was selected as the aerobic exercise of focus for this treatment because it is recommended for patients with all levels of pain severity, is highly feasible to complete, and has shown effects on outcomes such as pain and disability.
  Pro-Diary monitor: Participants will wear during 5 separate 7-day "home monitoring" periods to assess physical activity (objectively measured via accelerometry), and ecological momentary assessment (EMA) of mental and physical symptoms. EMA will be collected during Weeks 1, 6, 15, 24 and 36.
- Run-in Period: Baseline visit to T2 visit. Pre-treatment with exposure to the PainGuide website platform.
  PainGuide: A 4-week, online, self-management program for pain known as PainGuide (online or smart phone). Participants will use this during the run-in period as well as after the run-in period.
- Follow-up: This includes participants who are on follow-up due to one or more of the following reasons: Missed study visit timepoint (T2), On Follow-up/PGIC=1 at T2 or T3 visit, or post-treatment follow from T4 to T5 visit.
Period: T1 - Pre-Randomization: PainGuide run-in
Arm/Group | MBSR (mindfulness-based stress reduction) | PT and exercise | Acupressure | Duloxetine | Run-in Period | Follow-up
Started (Enrolled participants (T1)) | 0 | 0 | 0 | 0 | 494 | 0
Completed (Completed Run-in period and still on-study.) | 0 | 0 | 0 | 0 | 417 | 0
Not Completed | 0 | 0 | 0 | 0 | 77 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 35 | 0
Not completed — Screen Failure | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 37 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 3 | 0
Period: T2 (Randomization) - T3
Arm/Group | MBSR (mindfulness-based stress reduction) | PT and exercise | Acupressure | Duloxetine | Run-in Period | Follow-up
Started (Participants on-study at T2.) | 102 | 102 | 102 | 96 | 0 | 15
Attended Study Visit (Participants who attended T2 visit.) | 102 | 102 | 102 | 96 | 0 | 3
Completed (Of those who attended T2 visit, participants who attended T3.) | 79 | 90 | 79 | 83 | 0 | 2
Not Completed | 23 | 12 | 23 | 13 | 0 | 13
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 7 | 0 | 7 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 11 | 8 | 11 | 7 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 2 | 1 | 0 | 0
Not completed — Missed Timepoint | 4 | 3 | 3 | 2 | 0 | 12
Period: T3 (Re-randomization) - T4
Arm/Group | MBSR (mindfulness-based stress reduction) | PT and exercise | Acupressure | Duloxetine | Run-in Period | Follow-up
Started (Participants on study at T3.) | 80 | 73 | 100 | 61 | 0 | 47
Attended Study Visit (Participants who attended T3 visit. Of note, there are participants that missed T2 but attended T3. This accounts for the difference in participants that completed T3/Period 2 and those that started T3/Period 3.) | 80 | 73 | 100 | 61 | 0 | 47
Completed (Of those who attended T3 visit, participants who attended T4.) | 56 | 60 | 81 | 49 | 0 | 21
Not Completed | 24 | 13 | 19 | 12 | 0 | 26
Not completed — Adverse Event | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 8 | 6 | 7 | 6 | 0 | 2
Not completed — Withdrawal by Subject | 11 | 5 | 10 | 3 | 0 | 1
Not completed — Physician Decision | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Missed Timepoint | 3 | 1 | 2 | 2 | 0 | 23
Period: T4 - T5 (Follow-Up)
Arm/Group | MBSR (mindfulness-based stress reduction) | PT and exercise | Acupressure | Duloxetine | Run-in Period | Follow-up
Started (Participants on-study at T4 visit.) | 0 | 0 | 0 | 0 | 0 | 304
Attended Study Visit (Participants who attended T4 visit. Of note, there are participants that missed T3 but attended T4. This accounts for the difference in participants that completed T4/Period 3 and those that started T4/Period 4.) | 0 | 0 | 0 | 0 | 0 | 277
Completed (Participants who attended T5 and final study visit.) | 0 | 0 | 0 | 0 | 0 | 274
Not Completed | 0 | 0 | 0 | 0 | 0 | 30
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 21
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 7
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: 402 participants were randomized to a treatment at T2, but no baseline data on 2 participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Acupressure | PT and Exercise | MBSR (Mindfulness-based Stress Reduction) | Duloxetine | Total
Number analyzed (Participants) | 101 | 102 | 101 | 96 | 400
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 93 | 79 | 93 | 84 | 349
  >=65 years | 8 | 23 | 8 | 12 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] — Collected through Qualtrics administered survey
  years | 49.0 (11.9) | 51.0 (13.3) | 50.2 (10.7) | 50.0 (11.0) | 50.2 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 68 | 72 | 63 | 273
  Male | 31 | 34 | 29 | 33 | 127
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 6 | 5 | 6 | 26
  Not Hispanic or Latino | 86 | 87 | 87 | 85 | 345
  Unknown or Not Reported | 6 | 9 | 9 | 5 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 0 | 2
  Asian | 11 | 3 | 10 | 16 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 23 | 22 | 16 | 27 | 88
  White | 54 | 66 | 64 | 44 | 228
  More than one race | 6 | 7 | 6 | 7 | 26
  Unknown or Not Reported | 6 | 4 | 4 | 2 | 16
Region of Enrollment [Number; unit: participants]
  United States | 101 | 102 | 101 | 96 | 400
Education [Count of Participants; unit: Participants]
  Primary (Elementary School) | 0 | 0 | 0 | 0 | 0
  Lower Secondary (Middle School) | 0 | 0 | 0 | 1 | 1
  Upper Secondary (High School) | 3 | 4 | 5 | 3 | 15
  Diploma or equivalent (GED) | 9 | 5 | 4 | 8 | 26
  Some College/ Certificate | 26 | 36 | 28 | 19 | 109
  Vocational/Trade School | 6 | 6 | 6 | 4 | 22
  Bachelor's degree | 22 | 22 | 23 | 20 | 87
  Some Graduate or Professional School | 6 | 4 | 11 | 3 | 24
  Graduate or Professional School diploma | 28 | 25 | 24 | 38 | 115
  Unknown | 1 | 0 | 0 | 0 | 1
Employment Status [Count of Participants; unit: Participants]
  Full-time employment | 46 | 40 | 45 | 43 | 174
  Part-time employment | 16 | 12 | 14 | 17 | 59
  Not employed | 18 | 20 | 21 | 21 | 80
  Retired | 19 | 30 | 21 | 15 | 85
  Unknown | 2 | 0 | 0 | 0 | 2
Relationship Status [Count of Participants; unit: Participants]
  Divorced | 24 | 18 | 19 | 14 | 75
  Married | 48 | 47 | 55 | 55 | 205
  Never married | 21 | 31 | 23 | 18 | 93
  Separated | 3 | 1 | 1 | 3 | 8
  Widowed | 4 | 5 | 3 | 6 | 18
  Unknown | 1 | 0 | 0 | 0 | 1
Pain Duration [Mean (Standard Deviation); unit: months] — Population: Pain duration was unknown on 3 participants in the Acupressure arm and 1 participant in the PT arm. This question was not required, so patients could choose not to answer. This is reflected in the number analyzed category.
  months
    number analyzed (Participants) | 98 | 101 | 101 | 96 | 396
    (all) | 113 (155) | 133 (216) | 126 (183) | 145 (418) | 129 (262)
Annual Household Income [Count of Participants; unit: Participants]
  Less than $10,000 | 4 | 7 | 5 | 9 | 25
  $10,000 - $24,999 | 12 | 15 | 12 | 9 | 48
  $25,000 - $34,999 | 8 | 12 | 10 | 3 | 33
  $35,000 - $49,999 | 15 | 14 | 9 | 9 | 47
  $50,000 - $74,999 | 16 | 11 | 13 | 10 | 50
  $75,000 - $99,999 | 9 | 5 | 12 | 7 | 33
  $100,000 - $149,999 | 14 | 11 | 12 | 13 | 50
  $150,000 - $199,999 | 5 | 5 | 9 | 9 | 28
  $200,000 or more | 4 | 5 | 4 | 11 | 24
  Prefer not to answer | 12 | 16 | 14 | 16 | 58
  Unknown | 2 | 1 | 1 | 0 | 4
PROMIS Pain Interference [Mean (Standard Deviation); unit: units on a scale] — The PROMIS pain interference consists of 4 questions on a Likert scale ranging from 'Not at all" (1) to "Very much" (5). Total scores are between 4 and 20, with higher scores indicating increased pain interference. Population: Pain Interference was unknown on 3 participants in the Acupressure arm, 1 participant in the PT arm, 1 participant in the MBSR arm, and 1 participant in the Duloxetine arm. This question was not required, so patients could choose not to answer. This is reflected in the number analyzed category.
  units on a scale
    number analyzed (Participants) | 98 | 101 | 100 | 95 | 394
    (all) | 14.8 (3.2) | 14.9 (3.5) | 15.5 (3.0) | 14.8 (3.4) | 15.0 (3.3)
Pain, Enjoyment of Life, and General Activity (PEG) [Mean (Standard Deviation); unit: units on a scale] — This is a 3 question scale where participants select a between 0 (no pain) to 10 (pain is bad and completely interferes). Higher the scores the worse the pain. Population: PEG was unknown on 3 participants in the Acupressure arm, 1 participant in the PT arm, 1 participant in the MBSR arm, and 1 participant in the Duloxetine arm. This question was not required, so patients could choose not to answer. This is reflected in the number analyzed category.
  units on a scale
    number analyzed (Participants) | 98 | 101 | 100 | 95 | 394
    (all) | 6.4 (1.8) | 6.4 (1.9) | 6.6 (1.5) | 6.4 (1.9) | 6.4 (1.8)
PROMIS Physical Function [Mean (Standard Deviation); unit: units on a scale] — The PROMIS physical function consists of 3 questions on a Likert scale ranging from 'Unable to Do" (1) to "Without any difficulty" (5) and 2 questions on a Likert scale ranging from "Cannot Do" to "Not at all". Total scores are between 6 and 30, with higher scores indicating increased physical function. Population: PROMIS Physical Function was unknown on 3 participants in the Acupressure arm, 1 participant in the PT arm, 1 participant in the MBSR arm, and 2 participant in the Duloxetine arm. This question was not required, so patients could choose not to answer. This is reflected in the number analyzed category.
  units on a scale
    number analyzed (Participants) | 98 | 101 | 100 | 94 | 393
    (all) | 17.5 (4.7) | 17.3 (4.9) | 16.8 (4.1) | 17.8 (5.3) | 17.3 (4.7)
PROMIS Sleep Disturbance [Mean (Standard Deviation); unit: units on a scale] — The PROMIS sleep disturbance consists of 5 questions on a Likert scale ranging from 'Not at all" (1) to "Very much" (5) and 1 question on a Likert scale ranging from 'Very good' (1) to 'Very poor' (5). Total scores are between 6 and 30, with higher scores indicating increased sleep disturbance. Population: PROMIS Sleep Disturbance was unknown on 3 participants in the Acupressure arm, 2 participant in the PT arm, 1 participant in the MBSR arm, and 1 participant in the Duloxetine arm. This question was not required, so patients could choose not to answer. This is reflected in the number analyzed category.
  units on a scale
    number analyzed (Participants) | 98 | 100 | 100 | 95 | 393
    (all) | 19.4 (5.2) | 19.4 (5.6) | 19.1 (5.8) | 20.2 (5.4) | 19.5 (5.5)
PROMIS Depression [Mean (Standard Deviation); unit: units on a scale] — The PROMIS depression consists of 4 questions on a Likert scale ranging from 'Never' (1) to 'Always' (5). Total scores are between 4 and 20, with higher scores indicating increased depression. Population: PROMIS Depression was unknown on 4 participants in the Acupressure arm, 1 participant in the PT arm, 1 participant in the MBSR arm, and 2 participants in the Duloxetine arm. This question was not required, so patients could choose not to answer. This is reflected in the number analyzed category.
  units on a scale
    number analyzed (Participants) | 97 | 101 | 100 | 94 | 392
    (all) | 8.6 (4.3) | 8.1 (3.9) | 8.3 (3.8) | 7.8 (3.8) | 8.2 (3.9)
PROMIS Anxiety [Mean (Standard Deviation); unit: units on a scale] — The PROMIS anxiety consists of 4 questions on a Likert scale ranging from 'Never' (1) to "Always" (5). Total scores are between 4 and 20, with higher scores indicating increased anxiety. Population: PROMIS Anxiety was unknown on 4 participants in the Acupressure arm, 1 participant in the PT arm, 1 participant in the MBSR arm, and 2 participants in the Duloxetine arm. This question was not required, so patients could choose not to answer. This is reflected in the number analyzed category.
  units on a scale
    number analyzed (Participants) | 97 | 101 | 100 | 94 | 392
    (all) | 8.6 (4.2) | 7.7 (3.5) | 8.0 (3.5) | 8.0 (4.1) | 8.1 (3.8)
PROMIS Fatigue [Mean (Standard Deviation); unit: units on a scale] — The PROMIS fatigue consists of 4 questions on a Likert scale ranging from 'Not at all" (1) to "Very much" (5). Total scores are between 4 and 20, with higher scores indicating increased fatigue. Population: PROMIS Fatigue was unknown on 4 participants in the Acupressure arm, 1 participant in the PT arm, 3 participants in the MBSR arm, and 2 participants in the Duloxetine arm. This question was not required, so patients could choose not to answer. This is reflected in the number analyzed category.
  units on a scale
    number analyzed (Participants) | 97 | 101 | 98 | 94 | 390
    (all) | 12.9 (4.6) | 12.3 (4.5) | 12.3 (4.4) | 11.9 (4.6) | 12.3 (4.5)
PROMIS Social Roles and Activities [Mean (Standard Deviation); unit: units on a scale] — The PROMIS Social Roles and Activities consists of 4 questions on a Likert scale ranging from 'Always" (1) to "Never" (5). Total scores are between 4 and 20, with higher scores indicating increased ability to participate in social activities. Population: Pain Interference was unknown on 4 participants in the Acupressure arm, 1 participant in the PT arm, 3 participants in the MBSR arm, and 2 participants in the Duloxetine arm. This question was not required, so patients could choose not to answer. This is reflected in the number analyzed category.
  units on a scale
    number analyzed (Participants) | 97 | 101 | 98 | 94 | 390
    (all) | 11.3 (3.5) | 11.4 (3.9) | 11.3 (3.6) | 11.7 (4.1) | 11.4 (3.8)
PROMIS Cognitive Function [Mean (Standard Deviation); unit: units on a scale] — The PROMIS cognitive function consists of 2 questions on a Likert scale ranging from 'Not at all" (1) to "Very much" (5). Total scores are between 2 and 10, with higher scores indicating increased cognitive function. Population: PROMIS Cognitive Function was unknown on 4 participants in the Acupressure arm, 1 participant in the PT arm, 4 participants in the MBSR arm, and 2 participants in the Duloxetine arm. This question was not required, so patients could choose not to answer. This is reflected in the number analyzed category.
  units on a scale
    number analyzed (Participants) | 97 | 101 | 97 | 94 | 389
    (all) | 7.1 (1.9) | 7.2 (1.9) | 7.3 (2.0) | 7.2 (2.3) | 7.2 (2.0)
PROMIS Pain Intensity [Mean (Standard Deviation); unit: units on a scale] — The PROMIS pain intensity consists of 1 question on a Likert scale ranging from 'No Pain" (0) to "Worst Imaginable Pain" (10). Total scores are between 0 and 10, with higher scores indicating increased pain intensity. Population: PROMIS Pain Intensity was unknown on 3 participants in the Acupressure arm, 1 participant in the PT arm, 3 participants in the MBSR arm, and 2 participants in the Duloxetine arm. This question was not required, so patients could choose not to answer. This is reflected in the number analyzed category.
  units on a scale
    number analyzed (Participants) | 97 | 101 | 98 | 94 | 390
    (all) | 6.1 (1.6) | 6.4 (1.7) | 6.4 (1.5) | 6.3 (1.9) | 6.3 (1.7)
Michigan Body Map [Mean (Standard Deviation); unit: number of regions] — The Michigan Body Map is assessed electronically and assesses number of regions the study participant has pain, 0 (No Chronic Pain) - 36 (All Pain Regions). Population: The Michigan Body Map was unknown on 4 participants in the Acupressure arm, 1 participant in the PT arm, 2 participants in the MBSR arm, and 2 participants in the duloxetine arm. This question was not required, so patients could choose not to answer. This is reflected in the number analyzed category.
  number of regions
    number analyzed (Participants) | 97 | 101 | 99 | 94 | 391
    (all) | 8.8 (6.3) | 8.3 (6.3) | 8.7 (6.4) | 8.1 (6.6) | 8.5 (6.4)
Fibromyalgia Criteria [Count of Participants; unit: Participants] — Participants meeting the 2016 Fibromyalgia Criteria.
  1. Widespread pain index (WPI) and symptom severity score (SSS)
     WPI ≥ 7 and SSS ≥ 5 OR WPI 4-6 and SSS ≥ 9
  2. Generalized pain: pain in 4/5 regions
  3. Symptoms present ≥ 3 months Population: 2016 Fibromyalgia Criteria was unknown on 4 participants in the Acupressure arm, 1 participant in the PT arm, 3 participants in the MBSR arm, and 2 participants in the Duloxetine arm. This question was not required, so patients could choose not to answer. This is reflected in the number analyzed category.
  Participants
    number analyzed (Participants) | 97 | 101 | 98 | 94 | 390
    (all) | 17 | 21 | 20 | 20 | 78
PainDetect [Mean (Standard Deviation); unit: units on a scale] — The PainDetect measure consists of 14 questions - 7 questions on a Likert scale ranging from 'Never" (0) to "Very strongly" (5), 2 body region questions, 1 y/n question assessing pain, 1 visual question assessing type of back pain, and 3 questions on a Likert scale ranging from "none" (0) to "Max" (10). Higher scores indicating increase back pain in more regions. Population: PainDetect was unknown on 4 participants in the Acupressure arm, 5 participants in the PT arm, 5 participants in the MBSR arm, and 6 participants in the Duloxetine arm. This question was not required, so patients could choose not to answer. This is reflected in the number analyzed category.
  units on a scale
    number analyzed (Participants) | 97 | 97 | 96 | 90 | 380
    (all) | 11.3 (7.3) | 10.9 (6.9) | 11.8 (7.7) | 11.8 (8.1) | 11.5 (7.5)
General Sensitivity Scale (GSS-8) [Mean (Standard Deviation); unit: units on a scale] — GSS-8 measures sensitivity with 8 questions in a yes/no format. Scores range from 0 to 8 with higher scores indicating increased sensitivity.
  units on a scale | 2.0 (2.1) | 2.0 (1.9) | 1.7 (1.9) | 1.7 (1.9) | 1.9 (2.0)
Pain Catastrophizing Scale (PCS) [Mean (Standard Deviation); unit: units on a scale] — The Pain Catastrophizing Questionnaire consists of 13 questions on a Likert scale ranging from 'Not at all" (0) to "All the time" (4). Total scores are between 0 and 52, with higher scores indicating increased catastrophizing. Population: Pain Catastrophizing Scale (PCS) was unknown on 4 participants in the Acupressure arm, 1 participant in the PT arm, 1 participant in the MBSR arm, and 1 participant in the Duloxetine arm. This question was not required, so patients could choose not to answer. This is reflected in the number analyzed category.
  units on a scale
    number analyzed (Participants) | 97 | 101 | 100 | 95 | 393
    (all) | 12.4 (5.3) | 11.5 (5.7) | 12.0 (5.0) | 12.1 (6.2) | 12.0 (5.6)
Pain Self Efficacy Questionnaire (PSEQ) [Mean (Standard Deviation); unit: units on a scale] — The Pain Self Efficacy Quesionnaire (PSEQ) consists of 10 questions on a Likert scale ranging from 'Not at all confident" (0) to "Completely Confident" (6). Total scores are between 0 and 60, with higher scores indicating increased self efficacy. Population: Pain Self Efficacy Questionnaire (PSEQ) was unknown on 4 participants in the Acupressure arm, 2 participants in the PT arm, 3 participants in the MBSR arm, and 2 participants in the Duloxetine arm. This question was not required, so patients could choose not to answer. This is reflected in the number analyzed category.
  units on a scale
    number analyzed (Participants) | 97 | 100 | 98 | 94 | 389
    (all) | 6.9 (3.0) | 7.3 (3.2) | 7.0 (3.0) | 7.3 (3.0) | 7.1 (3.1)
Fear Avoidance Belief Questionnaire (FAPQ) [Mean (Standard Deviation); unit: units on a scale] — The Fear Avoidance Belief Questionnaire consists of 16 questions on a Likert scale ranging from 'Completely Disagree" (0) to "Completely Agree" (6). Total scores are between 0 and 96, with higher scores indicating fear avoidance. Population: Fear Avoidance Belief Questionnaire (FABQ) was unknown on 4 participants in the Acupressure arm, 2 participants in the PT arm, 5 participants in the MBSR arm, and 3 participants in the Duloxetine arm. This question was not required, so patients could choose not to answer. This is reflected in the number analyzed category.
  units on a scale
    number analyzed (Participants) | 97 | 100 | 96 | 93 | 386
    (all) | 15.1 (4.9) | 15.4 (4.9) | 15.9 (4.3) | 15.6 (5.3) | 15.5 (4.9)
Chronic Pain Acceptance Questionnaire (CPAQ) [Mean (Standard Deviation); unit: units on a scale] — The Chronic Pain Acceptance Questionnaire consists of 8 questions on a Likert scale ranging from 'Never" (0) to "Always true" (6). Total scores are between 0 and 48, with higher scores indicating increased pain acceptance. Population: Chronic Pain Acceptance Questionnaire (CPAQ) was unknown on 4 participants in the Acupressure arm, 2 participants in the PT arm, 6 participants in the MBSR arm, and 2 participants in the Duloxetine arm. This question was not required, so patients could choose not to answer. This is reflected in the number analyzed category.
  units on a scale
    number analyzed (Participants) | 97 | 100 | 95 | 94 | 386
    (all) | 24.2 (7.5) | 24.6 (7.8) | 24.0 (8.0) | 24.1 (7.1) | 24.2 (7.6)
Experiences Questionnaire (EQ-11) [Mean (Standard Deviation); unit: units on a scale] — The Experiences Questionnaire (EQ-11) consists of 11 questions on a Likert scale ranging from 'Never' (1) to 'All the time' (5). Total scores are between 11 and 55. A higher total score indicates a greater ability to decenter, which is a positive indicator of detached observation of one's internal experiences. Population: Experiences Questionnaire was unknown on 5 participants in the Acupressure arm, 2 participants in the PT arm, 6 participants in the MBSR arm, and 4 participants in the Duloxetine arm. This question was not required, so patients could choose not to answer. This is reflected in the number analyzed category.
  units on a scale
    number analyzed (Participants) | 94 | 100 | 95 | 92 | 381
    (all) | 39.1 (7.3) | 39.8 (7.5) | 38.9 (7.7) | 40.5 (7.4) | 39.6 (7.5)
Perceived Stress Scale (PSS) [Mean (Standard Deviation); unit: units on a scale] — The Perceived Stress Scale consists of 10 questions on a Likert scale ranging from 'Never' (0) to 'Very often' (4). Total scores are between 0 and 40, with higher scores indicating increased perceived stress. Population: Perceived Stress Scale was unknown on 4 participants in the Acupressure arm, 2 participants in the PT arm, 2 participants in the MBSR arm, and 3 participants in the Duloxetine arm. This question was not required, so patients could choose not to answer. This is reflected in the number analyzed category.
  units on a scale
    number analyzed (Participants) | 97 | 100 | 98 | 93 | 388
    (all) | 6.2 (3.4) | 5.8 (3.1) | 6.2 (3.4) | 6.0 (3.4) | 6.1 (3.3)
Positive and Negative Affect Scale (PANAS) [Mean (Standard Deviation); unit: units on a scale] — The Positive and Negative Affect Schedule (PANAS) is a 20-item self-report measure that assesses two distinct dimensions of mood: positive affect and negative affect. Participants rate the extent to which they have experienced each emotion over a specified time frame using a 5-point Likert scale - "Very slightly or not at all" (1) to "Extremely" (5). The PANAS score is separated into two subscales of Positive Affect (PA) and Negative Affect (NA), with a higher score indicating more positive or negative affect respectively. Each subscale ranges from 10-50. Population: Positive and Negative Affect Scale (PANAS) was unknown on 4 participants in the Acupressure arm, 2 participants in the PT arm, 5 participants in the MBSR arm, and 4/5 (positive/negative) participant in the Duloxetine arm. This question was not required, so patients could choose not to answer. This is reflected in the number analyzed category.
  units on a scale
    Positive Affect: number analyzed (Participants) | 97 | 100 | 96 | 92 | 385
    Positive Affect | 30.5 (8.1) | 31.0 (8.6) | 31.1 (8.0) | 31.6 (8.4) | 31.0 (8.3)
    Negative Affect: number analyzed (Participants) | 97 | 100 | 96 | 91 | 384
    Negative Affect | 21.3 (8.5) | 19.3 (7.1) | 20.3 (7.6) | 18.7 (7.5) | 19.9 (7.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference 4a Between Week 6 (T2) to Week 15 (T3)
Description: The PROMIS pain interference consists of 4 questions on a Likert scale ranging from 'Not at all" (1) to "Very much" (5). Total scores are between 4 and 20, with higher scores indicating increased pain interference.
Time Frame: week 6 (T2), week 15 (T3)
Population: Of the 402 participants who were randomized to a treatment, 331 who completed the T3 study visit were analyzed. Participants excluded from this analysis are those who did not complete either T2 or T3.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | MBSR (mindfulness-based stress reduction) | PT and exercise | Acupressure | Duloxetine
Number analyzed (Participants) | 79 | 90 | 79 | 83
score on a scale | -0.9 [-1.5 to -0.37] | -1.8 [-2.4 to -1.1] | -1.6 [-2.5 to -0.74] | -2.0 [-2.8 to -1.3]

2. Secondary Outcome: Change in the Pain, Enjoyment, and General Activity Scale (PEG) From Week 6 (T2) to Week 15 (T3)
Description: This is a 3 question scale where participants select a between 0 (no pain) to 10 (pain is bad and completely interferes). Higher the scores the worse the pain.
Time Frame: week 6 (T2), week 15 (T3)
Population: Of the 402 randomized participants, 331 who completed T3 study visit were analyzed. Participants excluded from this analysis are those who did not complete either T2 or T3.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Acupressure | PT and exercise | MBSR (mindfulness-based stress reduction) | Duloxetine
Number analyzed (Participants) | 79 | 90 | 79 | 83
score on a scale | -1.0 [-1.4 to -0.63] | -1.5 [-1.8 to -1.1] | -0.5 [-0.86 to -0.24] | -1.2 [-1.7 to -0.80]

3. Secondary Outcome: Patient Global Impression of Change (PGIC) From Week 6 (T2) to Week 15 (T3)
Description: This is a 1 question item where participants described their perceived improvement between T2 and T3 by selecting a score between 1 and 7, where 1 indicated "very much improved" and 7 indicated "very much worse. The lower the score, the greater improvement in perceived pain.
  Data is presented as count of participants who scored their improvement as a 1 or a 2 and those who scored their improvement as 3 or higher.
Time Frame: week 15 (T3)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | MBSR (mindfulness-based stress reduction) | PT and exercise | Acupressure | Duloxetine
Number analyzed (Participants) | 79 | 90 | 79 | 83
Participants
  Very much (score of 1) /much improved (score of 2) | 4 | 35 | 21 | 21
  Score 3 or higher | 75 | 55 | 58 | 62

ADVERSE EVENTS:
Time Frame: T1(Week 1) to T5 (Week 36), approximately 9 months
Description: In line with clinicaltrials.gov definitions.
Groups:
- Run-in Period: 5 week period leading up to randomization at T2 visit during which participants had access to the PainGuide self-managment program.
- On Follow-Up: Participants who were on follow-up due to PGIC=1 at T2 or T3, the week between treatment 1 and 2 or post treatment 2.
Arm/Group | MBSR (mindfulness-based stress reduction) | PT and exercise | Acupressure | Duloxetine | Run-in Period | On Follow-Up
All-Cause Mortality (participants affected / at risk) | 1/182 | 0/175 | 0/202 | 0/282 | 0/494 | 1/405
Serious Adverse Events (participants affected / at risk) | 5/182 | 8/175 | 6/202 | 3/167 | 9/494 | 17/405
Other Adverse Events (participants affected / at risk) | 1/182 | 1/175 | 0/202 | 40/282 | 4/494 | 2/405
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MBSR (mindfulness-based stress reduction) (N=182) | PT and exercise (N=175) | Acupressure (N=202) | Duloxetine (N=167) | Run-in Period (N=494) | On Follow-Up (N=405)
Chest Pain (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Breast Cancer (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Knee Replacement (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stroke (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
(General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Car Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous Cell Carcinoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pacemaker (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dizziness and Tingling Limbs (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nose Surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatomyositis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hernia Repair (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thrombectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Cardiac Seizure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Failure to Thrive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar Fusion (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DVT (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TKA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thyroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wrist Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Finger Surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hysterectomy (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TIA (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MBSR (mindfulness-based stress reduction) (N=182) | PT and exercise (N=175) | Acupressure (N=202) | Duloxetine (N=282) | Run-in Period (N=494) | On Follow-Up (N=405)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 13 (13) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 27 (27) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2025-09-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT04870957/Prot_000.pdf
  • Statistical Analysis Plan (2025-10-09): https://cdn.clinicaltrials.gov/large-docs/57/NCT04870957/SAP_001.pdf
  • Informed Consent Form (2025-01-30): https://cdn.clinicaltrials.gov/large-docs/57/NCT04870957/ICF_002.pdf